## Vernon Grant, PhD Assistant Research Professor Center for American Indian and Rural Health Equity Montana State University

NCT05314712

Document date: 01-06-25

## Study Protocol

**Objectives:** The objective of this 7-week sleep intervention is to increase nightly sleep in Blackfeet families with children in the K-3<sup>rd</sup> grade.

**Study Design:** The study was pre to post test nonrandomized trial of a 7-week sleep intervention.

Methods: We recruited 30 families of parent-child dyads to participate in a texting and Facebook child sleep intervention. Data was collected at 0 weeks and 8 weeks. Consent was sent to each family through email. Once consent was completed, they were instructed to report to the Blackfeet Tribal Council Chambers for data collection of height, weight, and demographic information. They were also administered four books from the Blackfeet Heritage Collection and given a cash incentive. It was up to each family to complete the surveys online that were sent through email. The following week began the 7-week sleep intervention. Each family was enrolled in a private Facebook page. Sleep strategies and Blackfeet language were sent to families in daily text messages. In the morning, Blackfeet prayers and common words were sent to participants. In the evening sleep strategies and book readings were sent to each family in an attempt to establish a bedtime routine. Many text messages were repeated and the content focused on turning off screens at least 1.5 hours before bedtime, establishing a relaxing bedtime routine, and waking up at the same time everyday. Facebook messages were posted about Blackfoot culture and songs. As with texts, this information was used to help establish a bedtime routine by listening to stories or singing songs in the Blackfoot culture. All correspondence were interactive, but participants rarely contacted our research team. At the conclusion of 7-weeks, survey data collection was repeated.

**IRB Approval:** This study was approved by the Blackfeet Nation Institutional Review Board.